CLINICAL TRIAL: NCT02530411
Title: A Randomised Double Blind Placebo Controlled Phase II Study of Fulvestrant With or Without the Addition of Vandetanib as Treatment for Patients With Metastatic Breast Cancer Resistant to Aromatase Inhibitor Therapy
Brief Title: Fulvestrant +/- Vandetanib in Advanced Aromatase Inhibitor Resistant Breast Cancer
Acronym: FURVA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Velindre NHS Trust (Other Government)
Collaborators: Cancer Research UK (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Lisette Nixon, Senior Trial Manager, Velindre NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014/VCC/0013; 2014-001208-23 (EudraCT Number)
Record Dates: First submitted 2015-03-23; First posted 2015-08-21 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Neoplasms
Keywords: Hormone resistance; vandetanib; fulvestrant
MeSH Terms: conditions — Neoplasms | interventions — Fulvestrant; vandetanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Fulvestrant 500mg Intra Muscular (IM) Day 1 (D1), D15, then D1 of every 28 day cycle Vandetanib 300 mg Per os (po) daily Clinician review D1, D15, weeks 4, 8, 12, 16, 20, 24 then 12 weekly. Computerised Axial Tomography (CT) at week 8, 16, 24 then 12 weekly.
  Interventions: Drug: Fulvestrant; Drug: Vandetanib
- Control (Placebo Comparator): Fulvestrant 500mg IM D1, D15, then D1 of every 28 day cycle Placebo po daily Clinician review D1, D15, weeks 4, 8, 12, 16, 20, 24 then 12 weekly. CT at week 8, 16, 24 then 12 weekly.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — The pharmacology and mode of action studies established that fulvestrant is the first agent in a new class of anti-estrogens that down-regulate the estrogen receptor (ER), and can therefore be described as an ER down-regulator.
  Other Names: FASLODEX™ (also previously known as ZD9238)
Drug: Vandetanib — Vandetanib is a potent inhibitor of the tyrosine kinase activity of vascular endothelial growth factor receptor (VEGFR; also known as kinase insert domain containing receptor)-2, an endothelial cell receptor for vascular endothelial growth factor (VEGF), and also possesses activity against epidermal growth factor receptor (EGFR) and Rearranged during Transfection (RET) tyrosine kinases.
  Other Names: CAPRELSA™ (also previously known as ZACTIMA™, ZD6474)
  Arms: Experimental

SUMMARY:
A randomised double blind placebo controlled phase II study of fulvestrant with or without the addition of vandetanib as treatment for patients with metastatic breast cancer resistant to aromatase inhibitor therapy.

DETAILED DESCRIPTION:
For patients with advanced breast cancer that has spread around the body, hormone therapy is often the best treatment. As well as being very effective, this means that patients do not experience the toxicity and inconvenience of chemotherapy. However, eventually the cancer is likely to become resistant to hormone therapy and in this situation, although other hormone drugs can be used, they sometimes do not work very well. So it is important to find ways of getting the cancer to respond to hormone treatment again.

There are many different ways in which breast cancer cells become resistant to hormone treatments, including a 'signalling' pathway in the cells called RET [Receptor tyrosine kinase RET] REarranged during Transfection. Research has shown increased activity of RET signalling pathways in hormone resistant cancer cells.

Vandetanib is an oral drug that inhibits RET signalling in cells and has been shown in laboratory studies to prevent the growth of breast cancer cells which have become resistant to hormone therapy. Hormone therapy drugs include tamoxifen, and the aromatase inhibitors (anastrozole, letrozole and exemestane). The investigators therefore believe that giving vandetanib together with hormone therapy may help prevent resistance to treatment in patients with breast cancer. In this trial the investigators will combine this drug with fulvestrant, another hormone therapy drug which is sometimes used alone in patients who have developed resistance to aromatase inhibitors, or tamoxifen. So patients entering the trial will have one drug, fulvestrant, which is known to work and may also be given the experimental drug, vandetanib.

To properly determine if vandetanib works as the investigators believe, this study will compare the activity of vandetanib combined with fulvestrant with fulvestrant combined with an inactive, 'placebo' tablet in a group of patients for whom treatment with single agent fulvestrant is thought appropriate. The investigators plan to recruit a total of 160 patients. Half of them will be given fulvestrant and vandetanib and half will be given fulvestrant and placebo, and the treatment a particular patient will get will be chosen by random chance. Neither the patient nor the patients doctor will know whether the patient is getting vandetanib or the inactive placebo. The most important measure of effect will be the time until the cancer grows again, but the study will also look closely at the side effects of the drugs. The investigators will also look at whether the way in which an individual responds relates to the results from laboratory studies on the RET pathways carried out on previously stored tumour samples. This will mean that patients will not need to have additional biopsy samples taken.

ELIGIBILITY:
Inclusion criteria:

1. Female ≥ 18 years
2. Post-menopausal
3. Minimum life expectancy 12 weeks
4. Histological confirmation of ER+ve breast cancer on primary tumour at diagnosis/on biopsy of metastasis
5. Histological confirmation of HER2 negative breast cancer on primary tumour at diagnosis/on biopsy of a metastasis
6. Clinical or histological confirmation of metastatic or locally advanced disease not amenable to curative surgical resection
7. ECOG 0-2 with no deterioration over previous 2 weeks
8. Measurable or non-measurable disease
9. Adequate bone marrow and organ function
10. Progressive disease whilst receiving third generation aromatase inhibitor for locally advanced or metastatic BC or relapsed with metastatic disease whilst receiving third generation AI in adjuvant setting
11. Radiological or objective clinical evidence of recurrence or progression on or after last systemic therapy prior to enrolment
12. ≤3 prior lines of endocrine therapy for ABC
13. ≤ 1 line of cytotoxic chemotherapy for ABC
14. Suitable for further endocrine therapy
15. Availability of archival tumour sample or fresh biopsy
16. Informed consent
17. Normal cardiac function

Exclusion criteria:

1. Previous treatment with fulvestrant or inhibitors of RET pathway
2. Last dose chemotherapy, immunotherapy targeted therapy, biological therapy or tumour embolisation <21 days (<6 weeks for nitrosurea or mitomycin C) prior to study treatment
3. Last dose of palliative radiotherapy <7 days prior to study treatment
4. Rapidly progressive visceral disease not suitable for further endocrine therapy
5. Spinal cord compression or brain/meningeal metastases unless asymptomatic, treated and stable and not requiring steroids for ≥ 4 weeks study treatment
6. Any of the following cardiac criteria: Significant cardiac event, superior vena cava syndrome, NYHA classification of heart disease ≥2 within 12 weeks before randomisation, or presence of cardiac disease that increases risk of ventricular arrhythmia; History of arrhythmia which is symptomatic or requires treatment, symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia; Congenital long QT syndrome; History of QT prolongation associated with other medications that required discontinuation of that medication; QTcB >480msec on screening ECG
7. Electrolyte values: Potassium <4.0 mmol/L despite supplementation, or above CTCAE Grade 1 upper limit, at randomisation; Magnesium below the normal range despite supplementation, or above CTCAE Grade 1 upper limit, at randomisation; Calcium (ionised or serum) below the normal range despite supplementation, or above Grade 1 upper limit, at randomisation
8. Creatinine clearance <30 ml/min. Patients with creatinine clearance <50 mL/min will start at a permanently reduced vandetanib dose of 200 mg.
9. Major surgery (excluding placement of vascular access) within 4 weeks before study treatment
10. Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C and HIV
11. With the exception of alopecia, any unresolved toxicities from previous therapy greater than CTCAE grade 1 before study treatment
12. Elevated ALP in absence of bone metastasis
13. History of hypersensitivity to active or inactive excipients of vandetanib or fulvestrant
14. Evidence of dementia, altered mental status or any psychiatric condition that would prohibit understanding or rendering of informed consent
15. Participation in another study with investigational product during last 30 days
16. Inability or unwillingness to comply with study procedures, including inability to take regular oral medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Time to event. This outcome will be assessed over an estimated period of up to 45 months.
  Time to event based on Response Evaluation Criteria in Solid Tumours (RECIST) v1.1. - Time from randomisation to any disease progression and/or death.

SECONDARY OUTCOMES:
Objective Response Rate | Time to event. This outcome will be assessed when all participants have completed a minimum 12 months follow-up and at least 98 disease progression events are observed, i.e. over an estimated period of up to 45 months.
  Objective Response Rate as assessed by the Response Evaluation Criteria in Solid Tumours (RECIST). Disease progression will be formally assessed according to the RECIST v1.1 criteria.
Overall Survival | Time to event. This outcome will be assessed over an estimated period of up to 45 months.
  Time from enrolment to death from any cause with those still alive censored at date last seen.
Exploratory analysis: The influence of RET signalling pathway components expression on vandetanib activity. | Data will be analysed when archival tumour tissue samples have been collected from all consenting patients. This outcome will be assessed and data presented up to 45 months.
  The influence of RET signalling pathway components expression on vandetanib activity.
Safety and tolerability of the fulvestrant/vandetanib trial drug regime measured by the number of participants with reported serious adverse events (composite outcome measure). | Initial safety reviews will be conducted after 20 and 40 patients have completed at least one cycle of treatment (estimated 8 and 16 months after enrolment of the first patient respectively). Final assessment/data presentation by 2018 (up to 45 months).
  This outcome will observe the number of side effects of the combined vandetanib and fulvestrant drug regime as recorded via real-time serious adverse event reporting.
Feasibility of use of the combined vandetanib/fulvestrant trial drug regime measured by the number of participants requiring dose delays, reductions and/or study withdrawal to manage reported serious adverse events. | Initial safety reviews will be conducted after 20 and 40 patients have completed at least one cycle of treatment (estimated 8 and 16 months after enrolment of the first patient respectively). Final assessment/data presentation by 2018 (up to 45 months).
  This outcome will assess the number of patients requiring dose delays, reductions, and/or study withdrawal to manage side effects recorded via real-time serious adverse event reporting.
Clinical Benefit Rate (measuring the proportion of patients with no disease progression after six months of treatment) | The trial data will be analysed when all participants have completed a minimum 12 months follow-up and at least 98 disease progression events are observed. This outcome will be assessed and the data presented up to 45 months.
  The clinical benefit rate will be assessed by measuring the proportion of patients with no disease progression after six months of treatment. Disease progression will be formally assessed according to the RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Beresford, MD MRCP FRCR, Study Director — Royal United Hospital NHS Trust, Bath, UK; Robert Jones, MD PhD MCRCP, Study Director — Velindre NHS Trust, Cardiff, UK
Locations (5):
- United Kingdom (5):
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Royal Devon and Exeter Hospital, Exeter, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Velindre Cancer Center, Velindre Hospital, Cardiff, Wales
  - Royal United Hospital Bath, Bath

REFERENCES:
- [Derived] Beresford M, Casbard A, Hudson Z, Carucci M, Ingarfield K, Gee J, Smith J, Kitson T, Alchami F, Madden TA, Hayward L, Hwang D, Spensley S, Waters S, Wheatley D, Jones RH. Fulvestrant plus vandetanib versus placebo for the treatment of patients with metastatic breast cancer resistant to aromatase inhibitor therapy (FURVA): a multicentre, Phase 2, randomised controlled trial. BJC Rep. 2023 Sep 14;1(1):13. doi: 10.1038/s44276-023-00016-8. PMID 39516358